CLINICAL TRIAL: NCT04464941
Title: Oral Health Promotion Program for Persons With Severe Mental Illness: A Cluster Randomized Controlled Study
Brief Title: Oral Health Promotion Program for Persons With Severe Mental Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Bing Show Chwan Memorial Hospital (Other)
Responsible Party: Principal Investigator, Po-Ren Teng, MD, PhD, Chang Bing Show Chwan Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RD103035018
Record Dates: First submitted 2020-07-07; First posted 2020-07-09 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Evaluate the Effects of an Oral Health Promotion Program
Keywords: oral health, promotion program, plaque index, mental illness
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Intervention Model Description: Cluster Randomized Controlled Study
Who Masked: Outcomes Assessor
Masking Description: Assessment of dental plaque was carried out by a single dentist, who was blind to group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- oral health promotion program (Experimental): The oral health promotion program was a composite intervention with both group and individual components. The group intervention consisted of:
  1. Group oral health education 2. Display of Bass tooth-brushing methods 3. Broadcasting of songs as tooth-brushing reminders; The individual interventions included:
  1. Instruction in the Bass tooth-brushing method 2. Individual behavioral modification method
  Interventions: Behavioral: a composite intervention with both group and individual components for oral health promotion program
- Usual care group (No Intervention)

INTERVENTIONS:
Behavioral: a composite intervention with both group and individual components for oral health promotion program — The group intervention consisted of:
  1. Group oral health education 2. Display of Bass tooth-brushing methods 3. Broadcasting of songs as tooth-brushing reminders; The individual interventions included:
  1. Instruction in the Bass tooth-brushing method, 2. Individual behavioral modification method
  Arms: oral health promotion program

SUMMARY:
A cluster randomized controlled study was carried out in chronic psychiatric wards of a general hospital in central Taiwan. Sixty-eight eligible male individuals admitted to 2 wards were randomly assigned to an experimental and a control group. Participants in the experimental group underwent an oral health promotion program that consisted of biweekly group education sessions, and a 12-week individual behavioral modification for oral hygiene course. The participants in the control group received usual care only. Dental plaque (measured by the Plaque Control Index) was examined by a single dentist before and after the experiment.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted in chronic psychiatric wards were eligible.

Exclusion Criteria:

* significant cognitive disabilities, severe hearing impairment, orthodontic appliances, an edentulous status, or a handicap when tooth-brushing

Ages: 20 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2016-03-21 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-07-10 (Actual)

PRIMARY OUTCOMES:
Dental Plaque Index | 12-week
  Plaque Control Index (PCI) developed by O'Leary et al. to score the primary outcome, plaque accumulation, on the surfaces of the teeth. The score was computed by the existence of plaque divided by all examined surfaces; a higher plaque index indicated poor oral hygiene. We calculated a person-level plaque score by averaging plaque scores for all teeth at each examination.

REFERENCES:
- [Derived] Kuo MW, Yeh SH, Chang HM, Teng PR. Effectiveness of oral health promotion program for persons with severe mental illness: a cluster randomized controlled study. BMC Oral Health. 2020 Oct 27;20(1):290. doi: 10.1186/s12903-020-01280-7. PMID 33109148